CLINICAL TRIAL: NCT05858073
Title: Immediate Effects of Kinesiotaping on Pain, Proprioception, and Posture in Round Shoulder Individuals With Subacromial Impingement Syndrome: A Double-Blinded Randomized Control
Brief Title: Investigation of Immediate Efficacy of Kinesiology Taping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-772.02-2825
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Postural; Defect
Keywords: taping

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping. (Other)
  Interventions: Other: Kinesio Taping
- Placebo Kinesio Taping. (Placebo Comparator)
  Interventions: Other: Placebo Kinesio Taping

INTERVENTIONS:
Other: Kinesio Taping — Standard 5 cm Kinesio Tex will be used. Initially, a Y-strip was paper-off (without tension) from the starting point to the insertion of the supraspinatus, while the participants were reaching with their upper extremities behind their backs and flexing their necks to the contralateral side. Second, an I-strip from the coracoid process will be applied around the posterior deltoid using approximately 50% to 75% downward flexion. Initially, the shoulder will be externally rotated without elevation, and then slightly horizontally adduction and forward elevation as the end of the band is applied without stretching. This I strip is shaped like a Y at the end of the tape.
  Finally, a Y-strip will be applied using paper-off tension from the T10-T12 region to the medial border of the scapula to facilitate the lower trapezius muscle. For this technique, the shoulder was adducted horizontally and the middle tail was applied with the hands crossed over the chest.
  Arms: Kinesio Taping.
Other: Placebo Kinesio Taping — Standard placebo taping will be applied to the placebo Kinesio taping group with a standard 5 cm Kinesio Tex. Two tension-free strips will be applied separately to the acromioclavicular joint and lower trapezius muscle. Suspicious participants will be excluded from the study.
  Arms: Placebo Kinesio Taping.

SUMMARY:
Shoulder protraction is the forward tilt of the head with hyperextension of the cervical spine and is associated with lengthening of the sternocleidomastoid and scalene muscles. With the lengthening of the flexor muscles, the weakened and shortened trapezius, levator scapula, and serratus anterior muscles lead to extra flexor torque and sustained contraction.

DETAILED DESCRIPTION:
Weakness in the rotator cuff muscles, especially infraspinatus and supraspinatus muscles, has been observed in individuals with scapular dyskinesia and who frequently use overhead movements in their daily lives. The most important point to be considered in the treatment of scapular dyskinesia is the effective evaluation and treatment of primary and secondary symptoms and conditions. The preference of shoulder rehabilitation programs in which the scapula is also included in the treatment program will provide great benefits to physiotherapists in terms of treatment. Effective treatment can be provided by taping, exercise and many other treatment methods.

ELIGIBILITY:
Inclusion Criteria:

* Those with neck pain
* Being between 18-60 years old

Exclusion Criteria:

* Hypertension
* Cardiopulmonary disease
* Pregnancy
* malignancy
* Operation, injection, etc. for the neck in the last 3 months. those with a history of treatment
* Spine surgery
* Psychological discomfort
* Neurological and orthopedic deficits

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | one day
  In the measurement of neck pain severity, it was planned to use a standard, proven 10 mm VAS. Patients will be asked to determine a value between 0 and 10 for the VAS, with 0 in the absence of pain and 10 mm in the most severe pain.
New York Posture Scale | one day
  Posture analysis is done while standing upright. Postures of the subjects participating in the study were evaluated with the New York Posture Scale. In this evaluation system, posture that can occur in 13 different parts of the body is evaluated. For scoring, a score of five was given if the person's posture was correct, three if it was moderately impaired, and one if it was severely impaired. The total score obtained with the test evaluation is a maximum of 65 and a minimum of 13. Standard evaluation criteria developed for this test were defined as "very good" if the total score was >=45, "good" if 40-44, "moderate" if 30-39, "poor" if 20-29, and "poor" if <=19. detected.
Proprioception Evaluation | one day
  An inclinometer is an instrument that records angular movements with respect to gravity. The inclinometer has many advantages such as precise measurement, digital display, and ease of use. In our study, inclinometer will be used to evaluate proprioception.
  The patient is first brought to 30° shoulder flexion position 3 times while standing and asked to memorize this position. Then the patient is asked to find the same position with his eyes closed. The patient is asked to return to the upright position and find the 30° flexion position. The same procedure is repeated in sitting position at 30° flexion and 15° extension positions. This process is repeated 3 times and the results are recorded. The average of these 3 measurements will be used in the analysis of the data.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçehir University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duperrat B, Puissant A, Larregue M, Fixy P. [Recklinghausen's neurofibromatosis with xanthoma]. Bull Soc Fr Dermatol Syphiligr. 1972;79(3):227. No abstract available. French. PMID 4629933
- [Derived] Demircioglu G, Genc H. Immediate effects of Kinesio taping on pain, proprioception, and posture in round shoulder individuals with subacromial impingement syndrome: A randomized, double-blinded controlled trial. Medicine (Baltimore). 2024 Dec 13;103(50):e40498. doi: 10.1097/MD.0000000000040498. PMID 39686459